CLINICAL TRIAL: NCT05387148
Title: The Efficacy and Neurobehavioural Mechanism of Cannabidiol (CBD) for Alcohol Dependence: An Exploratory Pilot Study
Brief Title: The Efficacy and Neurobehavioural Mechanism of Cannabidiol (CBD) for Alcohol Dependence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South West Sydney Local Health District (Other)
Collaborators: University of Sydney (Other); Lambert Initiative for Cannabinoid Therapeutics (Unknown)
Responsible Party: Principal Investigator, Kirsten Morley BPsych MPH PhD, Associate Professor Kirsten Morley, University of Sydney
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: X19-0416
Record Dates: First submitted 2022-05-15; First posted 2022-05-24 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol Withdrawal; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): For a total of three days, so that both study participants and staff are blind to treatment condition
  Interventions: Drug: Cannabidiol (CBD)
- Placebo (Placebo Comparator): For a total of three days, so that both study participants and staff are blind to treatment condition
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) — Four 200mg soft gel capsules of Cannabidiol (CBD) will be taken orally daily for a total of 3 days.
  Arms: Cannabidiol (CBD)
Drug: Placebo — The placebo will be identical in appearance, taste, and composition except for the active ingredient of pure CBD. So, four 200mg soft gel capsules of the placebo will be taken orally daily for a total of 3 days.
  Arms: Placebo

SUMMARY:
The study will explore the psychophysiological and neurobiological and mechanisms of CBD in participants with alcohol use disorder

DETAILED DESCRIPTION:
New treatment strategies for treating symptoms of alcohol dependence are urgently needed. Although alcohol related disorders are a leading cause of preventable death in Australia, their treatment is generally not evidence based. Cannabidiol (CBD) may serve as a novel pharmacotherapeutic due to its anxiolytic, anti-epileptic, neuro-protective, antioxidant and neuroprotective properties as well as a particularly safe side effect profile. Further, CBD has been shown to modulate drug craving and seeking behaviours.

This project will examine whether CBD exerts an effect on cue-induced craving by reducing activation in areas of the brain responsive to alcohol cues in comparison to a placebo. This study will use functional magnetic resonance imaging (fMRI) to examine activity in the brain while participants are exposed alcohol related cues and magnetic resonance spectroscopy (MRS) to determine levels of neurotransmitters that may be responsible for craving. In addition, we aim to investigate the effects of CBD on autonomic nervous system parameters associated with alcohol withdrawal symptoms and anxiety, such as heart rate variability and skin conductance. Additionally, clinical outcome measures will be taken to investigate CBDs influence on drinking, sleep

This project uses a randomised, double blind, crossover design with 800mg CBD vs matched placebo. The dosing paradigm will consist of one dose per day for three days per arm with a 18 days washout period in-between arms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages of 18 and 65 meeting DSM-5 criteria for current alcohol use disorder
* Adequate cognition and English language skills to give valid consent and complete research interviews;
* A BrAC reading of 0.00
* Must have a stable residence and be able to identify an individual who could locate subject if needed
* Provision of informed consent

Exclusion Criteria:

* Active major psychological disorder associated with psychosis, significant suicide risk
* Pregnancy or lactation - women shall be advised to use reliable contraception for the duration of drug therapy and a urine pregnancy test will be performed where necessary;
* Dependence on any substance other than nicotine (eg methadone)
* Diagnosis of epilepsy, and/or current use of anti-epileptic drugs (AED)
* Liver failure with jaundice or prolonged INR above 1.3
* Medical complications such as liver failure, cardiac ischemia or conduction abnormalities, renal impairment or unstable elevated vital signs (systolic blood pressure > 180, diastolic blood pressure > 120 or heart rate > 150)
* Severe cognitive impairment or insufficient English or literacy to complete study processes
* Concurrent use of drugs potentially exacerbated by CBD via CYP3A5 including cardiac medication (e.g. betablockers, calcium channel blockers and statins), macrolides and recent antihistamine use.
* Claustrophobia;
* Extreme obesity;
* Previous brain surgery;
* Ever employed as a machinist, a welder or a metal worker;
* Metal items such as pacemakers; aneurysm clips in the brain; metal dental implants; metallic fragments in the eye or anywhere else; insulin pump; metal implants; hearing aid or a prosthetic device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Changes in High Frequency Heart Rate Variability | 22 days
  To assess whether acute ingestion of CBD can modulate heart rate variability when responding to alcohol cues compared to neutral cues
Changes in Skin Conductance Levels | 22 days
  To assess whether acute ingestion of CBD modulates skin conductance levels when responding to alcohol cues compared to neutral cues
Changes in Brain Activation | 22 days
  To assess whether acute ingestion of CBD can attenuate brain activation via blood oxygen level dependent (BOLD) in areas associated with alcohol cue-elicited craving measured by an fMRI machine
Changes in Neurotransmitter levels in the Brain | 22 days
  To assess whether CBD treatment leads to changes in brain levels of the neurotransmitters: glutamate, gamma-aminobutyric acid (GABA), N-acetylaspartate (NAA) and glutathione (GSH)
Heavy Drinking Days | Up to 43 days
  Reduction in Heavy Drinking Days (HDD; defined as 4 or more drinks in a day for women and five or more drinks in a day for men). This will be measured by the Timeline Follow Back.
Absence of any Heavy Drinking Day | Up to 43 days
  Measured by Timeline Follow Back
Mean Alcohol Consumption per Drinking Day | Up to 43 days
  Measured by Timeline Follow Back
Alcohol Dependence Severity | Baseline
  Measured by the Alcohol Dependence Scale. The minimum score is 0 and the maximum score is 47. A higher score indicates more severe dependence.
Alcohol Craving | Up to 43 days
  As measured by the Penn Alcohol Craving Scale (PACS), which measures the amount of time spent thinking and craving for alcohol, difficulty in resisting consumption of alcohol if present and hypothetical pleasure associated with consumption of alcohol. This scale has a minimum score of 0 and a maximum score of 6. A higher score indicates greater levels of craving.

SECONDARY OUTCOMES:
Changes in Alcohol Craving | 22 days
  To assess whether acute ingestion of CBD can modulate subjective measures of alcohol cue elicited craving. This will be measured during the fMRI scan using the Visual Analogue Scale. This scale will assess alcohol craving, thirst and anxiety.
Changes in Alcohol Craving in response to alcohol cues | 22 days
  To assess whether acute ingestion of CBD can modulate subjective measures of alcohol cue elicited craving. This will be measured before and after the fMRI scan using the Alcohol Urge Questionnaire (AUQ). This Questionnaire consists of 8 questions that are scored on a Likert scale of 7 points. Two of the questions are reversed scored. Total score is computed by averaging the item scores. A greater score indicates greater craving.
Changes in Positive and Negative Mood States | 22 days
  To assess whether acute ingestion of CBD can modulate subjective measures of positive and negative mood states following alcohol cues. This will be measured before and after the fMRI scan using the Positive and Negative Affect Schedule (PANAS).
Changes in Anxiety | Up to 43 days
  Measured by cumulative scores on the DASS-21 Anxiety Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more anxiety.
Changes in Depression | Up to 43 days
  Measured by cumulative scores on the DASS-21 Depression Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates greater depression.
Changes in Stress | Up to 43 days
  Measured by cumulative scores on the DASS-21 Stress Scale. This scale has a minimum score of 0 and maximum score of 21. A higher score indicates more stress.
Sleep Disturbances | Up to 43 days
  As measured by the ISI (Insomnia Severity Index). This Index has a minimum score of 0 and a maximum score of 28. The higher the score indicates more severe insomnia.
Sleep Disturbances | 22 days
  To assess whether acute ingestion of CBD has any impact of sleep. This will be measured by an Actiwatch. The Actiwatch records motion and light to determine information about participants sleep and wake patterns. The participants will wear this watch for 48 hours on two separate occasions.
Changes in Tension Reduction Alcohol Expectancies | Up to 43 days
  To assess whether CBD treatment can reduce participants need to use alcohol to attenuate tension states (such as anxiety) as measured by the Tension Reduction subscale of the Alcohol Expectancy Questionnaire. Higher scores indicate greater reliance on alcohol to reduce tension/ anxiety.
Lifetime Consequences related to Drinking | Baseline
  To examine the adverse consequences a participant has experienced in their lifetime due to alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. This is measured using the Drinker Inventory of Consequences Lifetime Edition (DrInC-2L). Higher scores indicate more consequences.
Recent Consequences related to Drinking | Baseline
  To examine the adverse consequences a participant has experienced in the last 3 months due to alcohol abuse in five areas: Interpersonal, Physical, Social, Impulsive, and Intrapersonal. This is measured using the Drinker Inventory of Consequences Recent Edition (DrInC-2R). Higher scores indicate more consequences.
Behavioural Inhibition/Avoidance Scales | 22 days
  The BIS/BAS Scale is a 20-item self-report questionnaire designed to measure two motivational systems: the behavioral inhibition system (BIS), which corresponds to motivation to avoid aversive outcomes, and the behavioral activation system (BAS), which corresponds to motivation to approach goal-oriented outcomes.
Obsessive Compulsive Drinking | 22 days
  To assess an individuals obsessive thoughts about alcohol use and compulsive behaviours towards drinking as measured by the Obsessive Compulsive Drinking Scale. Six of the questions measure to obsession and eight of the questions measure compulsivity. Higher scores on these subscales indicate more obsession and compulsion, respectively.
Self-Confidence to Remain Abstinent | 22 days
  To measure an individual's self-confidence in avoiding alcohol through the Alcohol Abstinence Self-Efficacy Scale (AASE). There are 20 questions and each is scored from 0 to 4. Higher scores on this scale indicate more self-confidence.
Intolerance of Uncertainty | 22 days
  To assess an individual's reactions to situations that are ambiguous, the consequences of being uncertain, and attempts the individual might make to control the future. This will be measured through the Intolerance of Uncertainty Scale (IUS). This scale includes 27-items that are scored on a Likert scale (1 - Not at all characteristic of me to 5 - entirely characteristic of me). All scores are summed up and a higher score indicates greater inability to deal with uncertainty.
Impulsivity | 22 days
  To assess an individual's impulsivity across four domains: urgency, lack of premeditation and perseverance, and sensation seeking. This will be measured through the Impulsivity Scale (UPPS). Greater scores on this scale indicate greater impulsivity.
Alcohol Withdrawal | 22 days
  To assess an individual's severity of alcohol withdrawal through the Clinical Institute Withdrawal Assessment of Alcohol Scale - Revised (CIWA-Ar). Greater scores on this scale indicate the participant is experiencing greater alcohol withdrawal symptoms.
Approach and Avoidance towards Alcohol | Up to 43 days
  To assess an individual's automatic action tendencies (either approve or avoid) towards alcohol. This will be measured through the Approach Avoidance Task (AAT).
Response Time and Visuospatial Skills | Up to 43 days
  To assess an individual's response time and visuospatial skills through the Trail Making Test Part A (TMT-A).
Set-shifting Flexibility, Attention, and Inhibition | Up to 43 days
  To assess an individual's set-shifting flexibility, attention and inhibition through the Trail Making Test Part B (TMT-B).
Risk/Reward Taking Behaviour | Up to 43 days
  To assess an individual's risk taking behaviour measured through the Balloon Analogue Risk Task (BART).
Decision Making | Up to 43 days
  To assess an individual's decision making skills measured through the Columbia Card Task (CCT).
Response Inhibition | Up to 43 days
  To assess an individual's ability to inhibit prepotent responses measured through the Stroop task.
Working Memory Capacity to Update Information | Up to 43 days
  To assess an individual's capacity to update working memory information measured through the N-back task.
Working Memory Capacity to Shift Information | Up to 43 days
  To assess an individual's capacity to shift between two tasks measured by the Number Letter task.
Markers of neuroinflammation | Up to 43 days
  As measured by differences in blood sampling levels of glutathione.
Markers of Stress | Up to 43 days
  As measured by differences in blood sampling levels of cortisol. This will be measured at rest, before the fMRI scan and following the fMRI scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurzeler TP, Logge W, Watt J, DeMayo MM, Suraev A, McGregor IS, Haber PS, Morley KC. The neurobehavioural effects of cannabidiol in alcohol use disorder: Study protocol for a double-blind, randomised, cross over, placebo-controlled trial. Contemp Clin Trials Commun. 2024 Aug 13;41:101341. doi: 10.1016/j.conctc.2024.101341. eCollection 2024 Oct. PMID 39252861